CLINICAL TRIAL: NCT00426361
Title: A Multicentre Study to Evaluate the Immunogenicity and Safety of GSK Biologicals' HPV Vaccine (580299) Co-administered With Boostrix Polio (dTpa-IPV) in Healthy Female Subjects Aged 10-18 Years
Brief Title: Evaluation of Safety and Immunogenicity of Co-administering Human Papillomavirus (HPV) Vaccine With Other Vaccines in Healthy Female Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 108464
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Results first posted 2010-08-23 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2017-04

CONDITIONS: Infections, Papillomavirus
Keywords: Human Papillomavirus
MeSH Terms: conditions — Papillomavirus Infections | interventions — DTPa-HBV-IPV combined vaccine; halofantrine

ARMS (3):
- Cervarix Group (Experimental): Subjects who received GSK Biologicals' HPV-16/18 L1 AS04 vaccine (Cervarix TM) at Month 0, 1 and 6.
  Interventions: Biological: GSK Biologicals' HPV-16/18 L1 AS04 vaccine (Cervarix TM)
- Boostrix Polio → Cervarix Group (Experimental): Subjects who received Boostrix™ Polio at Month 0 and GSK Biologicals' HPV-16/18 L1 AS04 vaccine (Cervarix TM) at Month 1, 2 and 7.
  Interventions: Biological: Boostrix ® Polio; Biological: GSK Biologicals' HPV-16/18 L1 AS04 vaccine (Cervarix TM)
- Cervarix + Boostrix Polio Group (Experimental): Subjects who received GSK Biologicals' HPV-16/18 L1 AS04 vaccine (Cervarix TM) at Month 0, 1 and 6 with co-administration of Boostrix™ Polio at Month 0.
  Interventions: Biological: Boostrix ® Polio; Biological: GSK Biologicals' HPV-16/18 L1 AS04 vaccine (Cervarix TM)

INTERVENTIONS:
Biological: Boostrix ® Polio — One dose of vaccine administered intramuscularly
  Other Names: dTPa-IPV vaccine
  Arms: Boostrix Polio → Cervarix Group; Cervarix + Boostrix Polio Group
Biological: GSK Biologicals' HPV-16/18 L1 AS04 vaccine (Cervarix TM) — Three doses of vaccine administered intramuscularly, with the second and third dose give one month and six months after the first dose respectively
  Other Names: GlaxoSmithKline (GSK) Biologicals' HPV vaccine (580299); HPV-16/18 L1 AS04 vaccine

SUMMARY:
Infection with human papillomavirus (HPV) has been clearly established as the central cause of cervical cancer. Vaccination of pre-teens and adolescents, ideally before sexual debut and thus before exposure to oncogenic HPV, is a rational strategy for prevention of cervical cancer, and so HPV vaccination could complement the existing pre-adolescent/adolescents platform. Therefore, this Phase IIIb study is designed to evaluate the safety and immunogenicity of co-administering Boostrix polio (dTpa-IPV) with GSK Biologicals' (580299)HPV-16/18 L1 AS04 vaccine (Cervarix TM) as compared to the administration of either vaccine alone.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they and their parents/legally acceptable representatives can, and will, comply with the requirements of the protocol should be enrolled in the study.
* A female between, and including, 10 and 18 years of age at the time of the first vaccination.
* Written informed consent/assent obtained from the subject prior to enrolment. For subjects above the legal age of consent, written informed consent must be obtained from the subject. For subjects below legal age of consent, written informed consent obtained from the subject's parent/LAR, and written informed assent must be obtained from the subject.
* Healthy subjects, as established by medical history and history-directed physical examination, before entering into the study.
* Previously completed routine childhood vaccinations according to the recommended vaccination schedule at the time.
* Subjects must have a negative urine pregnancy test.
* Subject must be of non-childbearing potential, or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after completion of the vaccination series. Subjects who reach menarche during the study, and therefore become of childbearing potential, must agree to follow the same precautions.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period (up to Month 12/13).
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before and 30 days after each dose of vaccine(s). Administration of routine vaccines up to 8 days before the first dose of study vaccine is allowed. Enrolment will be deferred until the subject is outside of specified window.
* A woman planning to become pregnant, likely to become pregnant or planning to discontinue contraceptive precautions during the study period and up to two months after the last vaccine dose.
* Pregnant or breastfeeding women.
* Previous vaccination against HPV or planned administration of any HPV vaccine other than that foreseen by the study protocol during the study period.
* Previous administration of components of the investigational vaccine
* Administration of a diphtheria, tetanus, pertussis (DTP) vaccine, diphtheria-tetanus (Td) booster or dTpa vaccine within the previous five years.
* Administration of a pre-school booster of Oral Polio Vaccine (OPV) or Inactivated Polio Virus (IPV) vaccine (4 or 5th dose) within the previous five years.
* Hypersensitivity to latex.
* Known acute or chronic, clinically significant neurologic, hepatic or renal functional abnormality or thrombocytopenia, as determined by previous physical examination or laboratory tests.
* Cancer or autoimmune disease under treatment.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* History of encephalopathy within seven days of administration of a previous dose of pertussis vaccine that is not attributable to another identifiable cause.
* Temperature of >=40°C within 48 hours of receipt of a prior dose of DTP vaccine (DTPw and/or DTPa), not due to another identifiable cause.
* Collapse or shock-like state within 48 hours of receipt of a prior dose of DTP vaccine (DTPw and/or DTPa).
* Seizures with or without fever within three days of a prior dose of DTP vaccine (Diphtheria, Tetanus, whole cell Pertussis vaccine DTPw and/or Diphtheria, Tetanus, acellular Pertussis vaccine DTPa).
* Persistent, inconsolable crying lasting >=3 hours, occurring within 48 hours of a prior dose of DTP vaccine (DTPw and/or DTPa).
* Severe Arthus-type hypersensitivity reactions following a prior dose of tetanus toxoid within the previous 10 years.
* Known exposure to diphtheria or household exposure to pertussis within 30 days before (i.e., Day 0-29) vaccination with Diphtheria, Tetanus, acellular Pertussis and inactivated polio virus vaccine (dTpa-IPV).
* Diphtheria and/or tetanus and/or pertussis and/or polio diagnosed within 30 days before (i.e., Day 0-29) vaccination with dTpa-IPV.
* Presence of a contra-indication to vaccination according to the product leaflet of the commercially available dTpa-IPV vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period. Enrolment will be postponed until the subject is outside the specified window.

Ages: 10 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 751 (Actual)
Dates: Start 2007-02-13; Primary Completion 2008-03-17 (Actual); Study Completion 2008-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (33):
- France (14):
  - GSK Investigational Site, Auch
  - GSK Investigational Site, Draguignan
  - GSK Investigational Site, Essey-lès-Nancy
  - GSK Investigational Site, Évreux
  - GSK Investigational Site, Le Havre
  - GSK Investigational Site, Luynes
  - GSK Investigational Site, Montbrison
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pont-de-l'Arche
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Toulon
  - GSK Investigational Site, Tours
  - GSK Investigational Site, Vieux-Condé
- Germany (16):
  - GSK Investigational Site, Ettenheim, Baden-Wurttemberg
  - GSK Investigational Site, Karlsruhe, Baden-Wurttemberg
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Offenburg, Baden-Wurttemberg
  - GSK Investigational Site, Ravensburg, Baden-Wurttemberg
  - GSK Investigational Site, Rheinstetten, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Wolfenbüttel, Lower Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Nordhausen, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Spain (3):
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Seville

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Schwarz T et al. Co-administration of AS04-adjuvanted HPV-16/18 cervical cancer vaccine with DTPA-IPV in 10-18 year old girls: Month 7 results from a randomized trial. Abstract presented at the 27th annual ESPID meeting, Brussels, Belgium, 9-13 June 2009.
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- [Derived] Garcia-Sicilia J, Schwarz TF, Carmona A, Peters K, Malkin JE, Tran PM, Behre U, Iturbe EB, Catteau G, Thomas F, Dobbelaere K, Descamps D, Dubin G; HPV Vaccine Adolescent Study Investigators Network. Immunogenicity and safety of human papillomavirus-16/18 AS04-adjuvanted cervical cancer vaccine coadministered with combined diphtheria-tetanus-acellular pertussis-inactivated poliovirus vaccine to girls and young women. J Adolesc Health. 2010 Feb;46(2):142-51. doi: 10.1016/j.jadohealth.2009.11.205. PMID 20113920
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 108464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 108464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 108464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 108464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 108464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 108464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 108464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Cervarix Group: Subjects who received GSK Biologicals HPV 16/18 vaccine 580299 (CervarixTM) at Month 0, 1 and 6.
- Cervarix + Boostrix Polio Group: Subjects who received GSK Biologicals HPV 16/18 vaccine 580299 (CervarixTM) at Month 0, 1 and 6 with co-administration of Boostrix™ Polio at Month 0.
- Boostrix Polio → Cervarix Group: Subjects who received Boostrix™ Polio at Month 0 and GSK Biologicals HPV 16/18 vaccine 580299 (CervarixTM) at Month 1, 2 and 7.
Period: Overall Study
Arm/Group | Cervarix Group | Cervarix + Boostrix Polio Group | Boostrix Polio → Cervarix Group
Started | 248 | 255 | 248
Completed | 244 | 250 | 243
Not Completed | 4 | 5 | 5
Not completed — Lost to Follow-up | 3 | 2 | 5
Not completed — Withdrawal by Subject | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix Group | Cervarix + Boostrix Polio Group | Boostrix Polio → Cervarix Group | Total
Number analyzed (Participants) | 248 | 255 | 248 | 751
Age, Continuous [Mean (Standard Deviation); unit: years]
  Active phase (up to Month 7/8) | 13.9 (2.59) | 14.0 (2.43) | 13.9 (2.47) | 13.9 (2.50)
  Safety follow-up (up to Month 12/13) | 13.9 (2.58) | 13.9 (2.41) | 13.8 (2.46) | 13.9 (2.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 248 | 255 | 248 | 751
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Seroprotected Against Diphtheria and Tetanus
Description: Seroprotection against diphtheria and tetanus is defined as anti-diphtheria and anti-tetanus antibody titres greater than or equal to 0.1 International Units per Milliliter (≥ 0.1 IU/mL).
Time Frame: One month after vaccination with Boostrix Polio
Population: Analysis was performed on the Month 1 According-to-Protocol (ATP) cohort for analysis of immunogenicity and only on those subjects vaccinated with Boostrix Polio.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Cervarix + Boostrix Polio Group | Boostrix Polio → Cervarix Group
Number analyzed (Participants) | 0 | 240 | 233
Participants
  Diphtheria |  | 238 | 233
  Tetanus |  | 240 | 233

2. Primary Outcome: Titers of Anti-pertussis Toxoid (Anti-PT), Anti-pertactin Toxoid (Anti-PRN) and Anti-filamentous Hemagglutinin (Anti-FHA) Antibodies
Description: Titers are given as geometric mean titers (GMTs) calculated on all subjects and expressed as Enzyme-linked Immunosorbent Assay Units per Milliliter (EL.U/mL).
Time Frame: One month after vaccination with Boostrix Polio
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Group | Cervarix + Boostrix Polio Group | Boostrix Polio → Cervarix Group
Number analyzed (Participants) | 0 | 240 | 233
EL.U/mL
  Anti-PT: number analyzed (Participants) | 0 | 238 | 229
  Anti-PT |  | 84.2 [73.6 to 96.4] | 75.4 [65.6 to 86.8]
  Anti-FHA |  | 611.7 [553.6 to 675.9] | 615.2 [552.3 to 685.2]
  Anti-PRN: number analyzed (Participants) | 0 | 239 | 233
  Anti-PRN |  | 426.2 [368.1 to 493.4] | 360.0 [299.3 to 433.1]

3. Primary Outcome: Number of Subjects Seroprotected Against Poliovirus Type 1 (Polio 1), Polio 2 and Polio 3
Description: Seroprotection against polio 1, 2 and 3 is defined as anti-polio 1, 2 and 3 antibody titers greater than or equal to 8 Effective Dose 50% (≥ 8 ED50).
Time Frame: One month after vaccination with Boostrix Polio
Population: Analysis was performed on the Month 1 According-to-Protocol (ATP) cohort for analysis of immunogenicity and only on those subjects vaccinated with Boostrix Polio and with available results for the defined antigen.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Cervarix + Boostrix Polio Group | Boostrix Polio → Cervarix Group
Number analyzed (Participants) | 0 | 240 | 232
Participants
  Polio 1: number analyzed (Participants) | 0 | 240 | 231
  Polio 1 |  | 239 | 231
  Polio 2 |  | 240 | 232
  Polio 3: number analyzed (Participants) | 0 | 239 | 232
  Polio 3 |  | 239 | 232

4. Secondary Outcome: Number of Subjects Seroconverted for Anti-human Papilloma Virus 16 (Anti-HPV-16) and Anti-HPV-18 Antibodies After Completing the Cervarix Vaccination Course
Description: Seroconversion is defined as the appearance of antibodies with titers greater than or equal to the predefined cut-off value in the serum of subject seronegative before vaccination. Cut-off values assessed include 8 enzyme-linked immunosorbent assay units per milliliter (EL.U/mL) for anti-HPV-16 antibodies and 7 EL.U/mL for anti-HPV-18 antibodies.
Time Frame: One month post Cervarix Dose 3 (Month 7/8)
Population: Analysis was performed on the Month 7/8 According-to-Protocol (ATP) cohort for analysis of immunogenicity on subjects with available results for the defined antibody.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Cervarix + Boostrix Polio Group | Boostrix Polio → Cervarix Group
Number analyzed (Participants) | 198 | 204 | 204
Participants
  Anti-HPV-16: number analyzed (Participants) | 198 | 202 | 204
  Anti-HPV-16 | 198 | 201 | 204
  Anti-HPV-18: number analyzed (Participants) | 191 | 204 | 203
  Anti-HPV-18 | 191 | 203 | 203

5. Secondary Outcome: Number of Subjects Seroconverted for Anti-HPV-16 and Anti-HPV-18 Antibodies After Incomplete Cervarix Vaccination Course
Description: as for outcome 4
Time Frame: One month post Dose 1
Population: Analysis was performed on the Month 1 According-to-Protocol (ATP) cohort for analysis of immunogenicity and only on subjects from the Cervarix and Cervarix + Boostrix Polio groups with available results for the defined antibody.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Cervarix + Boostrix Polio Group | Boostrix Polio → Cervarix Group
Number analyzed (Participants) | 198 | 204 | 0
Participants
  Anti-HPV-16: number analyzed (Participants) | 198 | 202 | 0
  Anti-HPV-16 | 198 | 201 |
  Anti-HPV-18: number analyzed (Participants) | 191 | 204 | 0
  Anti-HPV-18 | 191 | 203 |

6. Secondary Outcome: Titers of Anti-human Papilloma Virus 16 (Anti-HPV-16) and Anti-human Papilloma Virus 18 (Anti-HPV-18) Antibodies After Completing the Cervarix Vaccination Course
Description: Titers are given as Geometric Mean Titers (GMTs) expressed as Enzyme-linked Immunosorbent Assay Units Per Milliliter (EL.U/mL).
Time Frame: One month post Cervarix Dose 3 (Month 7/8)]
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Group | Cervarix + Boostrix Polio Group | Boostrix Polio → Cervarix Group
Number analyzed (Participants) | 213 | 222 | 218
EL.U/mL
  Anti-HPV-16 | 18363.6 [16243.0 to 20761.0] | 15370.2 [13350.9 to 17694.8] | 14089.5 [12460.9 to 15930.9]
  Anti-HPV-18: number analyzed (Participants) | 210 | 218 | 216
  Anti-HPV-18 | 7032.8 [6220.7 to 7950.9] | 6630.4 [5768.0 to 7621.6] | 5135.0 [4537.3 to 5811.5]

7. Secondary Outcome: Titers of Anti-diphtheria and Anti-tetanus Antibodies
Description: Titers are given as Geometric Mean Titers (GMTs) and expressed as IU/mL.
Time Frame: One month after vaccination with Boostrix-Polio
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Cervarix Group | Cervarix + Boostrix Polio Group | Boostrix Polio → Cervarix Group
Number analyzed (Participants) | 0 | 240 | 233
IU/mL
  Anti-diphtheria |  | 5.085 [4.551 to 5.681] | 5.466 [4.896 to 6.103]
  Anti-tetanus |  | 8.552 [7.889 to 9.272] | 9.039 [8.321 to 9.818]

8. Secondary Outcome: Number of Subjects With Anti-diphtheria and Anti-tetanus Antibody Titers Above 1.0 International Units Per Milliliter (IU/mL)
Description: Anti-diphtheria and anti-tetanus antibodies cut-off value assessed include 1.0 IU/mL.
Time Frame: One month after vaccination with Boostrix Polio
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Cervarix + Boostrix Polio Group | Boostrix Polio → Cervarix Group
Number analyzed (Participants) | 0 | 240 | 233
Participants
  Anti-diphtheria |  | 231 | 226
  Anti-tetanus |  | 239 | 233

9. Secondary Outcome: Anti-poliovirus Type 1 (Anti-polio 1), Anti-polio 2 and Anti-polio 3 Antibody Titers
Description: Titers are given as Geometric Mean Titers (GMTs). The titer is a serum dilution giving 50 percent reduction of signal compared to control without serum.
Time Frame: One month after vaccination with Boostrix Polio
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cervarix Group | Cervarix + Boostrix Polio Group | Boostrix Polio → Cervarix Group
Number analyzed (Participants) | 0 | 240 | 232
titer
  Anti-polio 1: number analyzed (Participants) | 0 | 240 | 231
  Anti-polio 1 |  | 2045.1 [1714.7 to 2439.2] | 2390.5 [2021.4 to 2826.9]
  Anti-polio 2 |  | 2151.1 [1806.5 to 2561.6] | 2158.1 [1821.3 to 2557.1]
  Anti-polio 3: number analyzed (Participants) | 0 | 239 | 232
  Anti-polio 3 |  | 2777.2 [2376.5 to 3245.4] | 2732.5 [2318.0 to 3221.2]

10. Secondary Outcome: Number of Subjects With Booster Response to Diphtheria and Tetanus
Description: Booster responses to diphtheria and tetanus were defined as:
  * For initially seronegative subjects (pre-vaccination titer below cut-off value of 0.1 International Units per Milliliter): antibody titers at least four times the cut-off (post-vaccination titer greater than or equal to 0.4 IU/mL), and
  * For initially seropositive subjects (pre-vaccination titer greater than or equal to 0.1 IU/mL): an increase in antibody titers of at least four times the pre-vaccination titer.
Time Frame: One month after vaccination with Boostrix Polio
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Cervarix + Boostrix Polio Group | Boostrix Polio → Cervarix Group
Number analyzed (Participants) | 0 | 240 | 232
Participants
  Diphtheria |  | 160 | 159
  Tetanus |  | 167 | 161

11. Secondary Outcome: Number of Subjects With Booster Response to Pertussis Toxoid (PT), Pertactin Toxoid (PRN) and Filamentous Hemagglutinin (FHA)
Description: Booster response to PT, FHA and PRN were defined as:
  * For initially seronegative subjects [pre-vaccination titer below cut-off value of 5 enzyme-linked immunosorbent assay units per milliliter (EL.U/mL)]: antibody titers at least 4 times the cut-off,
  * For initially seropositive subjects with pre-vaccination titer above 5 EL.U/mL and < 20 EL.U/mL: an increase in antibody titers of at least 4 times the pre-vaccination titer,
  * For initially seropositive subjects with pre-vaccination titer above 20 EL.U/mL: an increase in antibody titers of at least 2 times the pre-vaccination titer.
Time Frame: One month after vaccination with Boostrix Polio
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Cervarix + Boostrix Polio Group | Boostrix Polio → Cervarix Group
Number analyzed (Participants) | 0 | 238 | 230
Participants
  PT: number analyzed (Participants) | 0 | 236 | 228
  PT |  | 199 | 182
  FHA: number analyzed (Participants) | 0 | 235 | 226
  FHA |  | 210 | 205
  PRN |  | 222 | 207

12. Secondary Outcome: Number of Subjects Reporting Solicited Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling at the injection site.
  Solicited general symptoms assessed include arthralgia, fatigue, fever (above 37.5 degree Celsius), gastrointestinal symptoms, headache, myalgia, rash and urticaria.
Time Frame: During the 7-day period (Day 0-6) following each vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, on subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Cervarix + Boostrix Polio Group | Boostrix Polio → Cervarix Group
Number analyzed (Participants) | 246 | 253 | 247
Participants
  Pain | 225 | 237 | 233
  Redness | 110 | 128 | 140
  Swelling | 124 | 125 | 123
  Arthralgia | 58 | 71 | 77
  Fatigue | 109 | 135 | 121
  Fever | 30 | 46 | 37
  Gastrointestinal symptoms | 51 | 63 | 61
  Headache | 111 | 138 | 122
  Myalgia | 107 | 144 | 127
  Rash | 20 | 27 | 17
  Urticaria | 12 | 11 | 15

13. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events
Description: Unsolicited adverse event = Any adverse event (AE) reported in addition to those solicited during the clinical study. Also any "solicited" symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event.
Time Frame: During the 30-day period (Day 0-29) following vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Cervarix + Boostrix Polio Group | Boostrix Polio → Cervarix Group
Number analyzed (Participants) | 248 | 255 | 248
Participants | 85 | 74 | 99

14. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events as New Onset Chronic Diseases (NOCDs) and Other Medically Significant Adverse Events (MSAEs)
Description: NOCDs assessed include e.g. autoimmune disorders, asthma, type I diabetes. MSAEs assessed include AEs prompting emergency room or physician visits that are not related to common diseases or SAEs that are not related to common diseases.
Time Frame: During the active phase of the study (up to Month 7/8) and during the safety follow-up (up to Month 12/13)
Population: Analysis was performed on the Total Vaccinated Cohort (for the active phase) and on the Extended Safety Follow-up Vaccinated Cohort (for the safety follow-up).
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Cervarix + Boostrix Polio Group | Boostrix Polio → Cervarix Group
Number analyzed (Participants) | 248 | 255 | 248
Participants
  NOCDs [Active phase] | 5 | 9 | 9
  NOCDs [Safety follow-up]: number analyzed (Participants) | 244 | 250 | 243
  NOCDs [Safety follow-up] | 0 | 0 | 0
  MSAEs [Active phase] | 35 | 27 | 49
  MSAEs [Safety follow-up]: number analyzed (Participants) | 244 | 250 | 243
  MSAEs [Safety follow-up] | 7 | 3 | 5

15. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: Serious adverse events assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: During the active phase of the study (up to Month 7/8) and during the safety follow-up (up to Month 12/13)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Cervarix + Boostrix Polio Group | Boostrix Polio → Cervarix Group
Number analyzed (Participants) | 248 | 255 | 248
Participants
  Active phase | 2 | 4 | 2
  Safety follow-up: number analyzed (Participants) | 244 | 250 | 243
  Safety follow-up | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: During the 7 day follow-up period after any vaccination for other (non-serious) adverse events. During the entire study period (12 months for Cervarix and Cervarix + Boostrix groups and 13 months for Cervarix → Boostrix group) for serious adverse events.
Description: For other (non-serious) adverse events collected by systematic assessment, the number of subjects at risk corresponds to the number of subjects from the Total Vaccinated Cohort with a documented dose.
Arm/Group | Cervarix Group | Cervarix + Boostrix Polio Group | Boostrix Polio → Cervarix Group
Serious Adverse Events (participants affected / at risk) | 3/248 | 4/255 | 3/248
Other Adverse Events (participants affected / at risk) | 232/248 | 245/255 | 242/248
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=248) | Cervarix + Boostrix Polio Group (N=255) | Boostrix Polio → Cervarix Group (N=248)
Appendicitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Imminent abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Tonsillitis streptococcal (Infections and infestations) | 0 | 0 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cervarix Group (N=248) | Cervarix + Boostrix Polio Group (N=255) | Boostrix Polio → Cervarix Group (N=248)
Pain (General disorders) | 225/246 | 237/253 | 233/247
Redness (General disorders) | 110/246 | 128/253 | 140/247
Swelling (General disorders) | 124/246 | 125/253 | 123/247
Arthralgia (General disorders) | 58/246 | 71/253 | 77/247
Fatigue (General disorders) | 109/246 | 135/253 | 121/247
Fever (above 37.5 degree Celsius) (General disorders) | 30/246 | 46/253 | 37/247
Gastrointestinal symptoms (General disorders) | 51/246 | 63/253 | 61/247
Headache (General disorders) | 111/246 | 138/253 | 122/247
Myalgia (General disorders) | 107/246 | 144/253 | 127/247
Rash (General disorders) | 20/246 | 27/253 | 17/247
Urticaria (General disorders) | 12/246 | 11/253 | 15/247
Upper respiratory tract infection (Infections and infestations) | 14 | 4 | 10
Headache (Nervous system disorders) | 4 | 6 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.